CLINICAL TRIAL: NCT02376816
Title: Phase I Gene Transfer Clinical Trial for Duchenne Muscular Dystrophy Using rAAVrh74.MCK.Micro-dystrophin
Brief Title: Clinical Intramuscular Gene Transfer Trial of rAAVrh74.MCK.Micro-Dystrophin to Patients With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jerry R. Mendell (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Jerry R. Mendell, Director, Center for Gene Therapy, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-00718
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; muscular dystrophy; dystrophin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: Low Dose (Experimental): The rAAVrh74.MCK.micro-Dystrophin vector will be injected to the Extensor Digitorum Brevis (EDB) muscle of a single foot at a total dose of 3E11 vg. The contralateral EDB muscle will injected with normal saline placebo as a comparator. Both physician and study team will be blinded as to which muscle received vector vs placebo. A minimum of three (3) patients with DMD will be enrolled in this cohort.
  Interventions: Biological: rAAVrh74.MCK.micro-Dystrophin
- Cohort 2: High Dose (Experimental): The rAAVrh74.MCK.micro-Dystrophin vector will be injected to the Extensor Digitorum Brevis (EDB) muscle of a single foot at a total dose of 1E12 vg. The contralateral EDB muscle will injected with normal saline placebo as a comparator. Both physician and study team will be blinded as to which muscle received vector vs placebo. A minimum of three (3) patients with DMD will be enrolled in this cohort.
  Interventions: Biological: rAAVrh74.MCK.micro-Dystrophin

INTERVENTIONS:
Biological: rAAVrh74.MCK.micro-Dystrophin — Recombinant adeno-associated virus carrying a truncated "micro" dystrophin transgene under control of a muscle specific MCK promoter.

SUMMARY:
The proposed phase I clinical trial is a pilot study to evaluate safety and biological activity of the rAAVrh74.MCK.micro-Dystrophin vector administered by an intramuscular route. This study will evaluated the micro-Dystrophin vector as a potential dystrophin replacement mechanism for Duchenne Muscular Dystrophy. Two cohorts will undergo gene transfer in a standard three-six dose escalation scheme to establish maximum tolerated dose (MTD) using toxicity. A minimum of three subjects will be enrolled into each cohort. The first cohort will receive a total dose of 3E11 vg. The second cohort will receive 1E12 vg total dose.

DETAILED DESCRIPTION:
The primary objective of this study is the assessment of the safety of an intramuscular administration of rAAVrh74.MCK.micro-Dystrophin to the Extensor Digitorum Brevis (EDB) muscle of patients with Duchenne Muscular Dystrophy (DMD). Safety will be assessed by changes in hematology, serum chemistry, urinalysis, immunologic response to rAAVrh74 and micro-Dystrophin protein, and reported history and observations of symptoms. Subjects will be evaluated at baseline, injection visit (days 0-2), and return for follow up visits on days 7, 14, 30,60, 90, and 180 and at the end of 1st and 2nd years. On Day 180, subjects will undergo a muscle biopsy on the injected muscles in one foot compared with placebo-treatment in the opposite foot to establish transgene expression and any potential toxicity from gene transfer.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 or older; must be wheelchair-dependent
* Confirmed Dystrophin mutations based on mutation compatibility with micro-dys cDNA based on previously published methods.
* Males of any ethnic group will be eligible.
* Ability to cooperate with muscle testing.
* Willingness of sexually active subjects with reproductive capacity to practice reliable method of contraception (If appropriate).

Exclusion Criteria:

* Active viral infection based on clinical observations.
* Symptoms or signs of cardiomyopathy, including:

  * Dyspnea on exertion, pedal edema, shortness of breath upon lying flat, or rales at the base of the lungs
  * Echocardiogram with ejection fraction below 40%
* Serological evidence of HIV infection, or Hepatitis A, B or C infection
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer.
* Subjects with AAVrh74 binding antibody titers ≥ 1:50 as determined by ELISA immunoassay.
* Abnormal laboratory values in the clinically significant range as defined in protocol or based upon normal values in the Nationwide Children's Hospital Laboratory.

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Safety based on number of participants with adverse events | 2 years
  AEs will be monitored and scored for severity and relatedness to the study article.

SECONDARY OUTCOMES:
Transgene Expression | 180 Days
  Biologic activity of the vector will be measured by immunohistochemistry detection of dystrophin on muscle biopsies as compared to placebo treated controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Mendell, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Rodino-Klapac LR, Montgomery CL, Mendell JR, Chicoine LG. AAV-mediated gene therapy to the isolated limb in rhesus macaques. Methods Mol Biol. 2011;709:287-98. doi: 10.1007/978-1-61737-982-6_19. PMID 21194036
- [Background] Rodino-Klapac LR, Montgomery CL, Bremer WG, Shontz KM, Malik V, Davis N, Sprinkle S, Campbell KJ, Sahenk Z, Clark KR, Walker CM, Mendell JR, Chicoine LG. Persistent expression of FLAG-tagged micro dystrophin in nonhuman primates following intramuscular and vascular delivery. Mol Ther. 2010 Jan;18(1):109-17. doi: 10.1038/mt.2009.254. Epub 2009 Nov 10. PMID 19904237
- [Background] Rodino-Klapac LR, Janssen PM, Montgomery CL, Coley BD, Chicoine LG, Clark KR, Mendell JR. A translational approach for limb vascular delivery of the micro-dystrophin gene without high volume or high pressure for treatment of Duchenne muscular dystrophy. J Transl Med. 2007 Sep 24;5:45. doi: 10.1186/1479-5876-5-45. PMID 17892583
- See also: Center for Gene Therapy, The Research Institute at Nationwide Children's Hospital — http://www.nationwidechildrens.org/center-for-gene-therapy
- See also: Senator Paul D. Wellstone Muscular Dystrophy Cooperative Research Center at Nationwide Children's Hospital — http://www.nationwidechildrens.org/wellstone-center
- See also: Gene Therapy Clinical Studies at Nationwide Children's Hospital — http://www.nationwidechildrens.org/gene-therapy-clinical-studies--1